CLINICAL TRIAL: NCT06782087
Title: A Comparative Study Between the Efficacy of Diode Laser and Nano-chitosan Gel on Activation of Non-vital in- Office Bleaching Agent :A Controlled Clinical Trial
Brief Title: A Comparative Study Between the Efficacy of Diode Laser and Nano-chitosan Gel on Activation of Non-vital in- Office Bleaching Agent
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Silvia Sabry, lecturer of conservative dentidtry, Misr University for Science and Technology
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022/0037
Record Dates: First submitted 2024-12-23; First posted 2025-01-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-05

CONDITIONS: Tooth Discoloration
Keywords: chitosan nanoparticles; Diode laser; carbamide peroxide; nonvital teeth bleaching
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- peroxides and sodium perborate and 980nm diode laser. (Other): peroxides and sodium perborate + 980nm diode laser.
  Interventions: Drug: nano chitosan

INTERVENTIONS:
Drug: nano chitosan — nano chitosan

SUMMARY:
The growing demand for white smile between patients has increased over recent years, the development of techniques and improvement of materials permits searching for beautiful natural smile.

The discoloration of teeth might be intrinsic, extrinsic, or combined. A variety of commercial bleaching agents is available. The most common substances used are carbamide peroxide or hydrogen peroxide or a mixture of sodium perborate and hydrogen peroxide.

DETAILED DESCRIPTION:
The aim of the study is to assess the effectiveness of two different in-office bleaching materials carbamide peroxide alone and carbamide peroxide with Chitosan nanoparticles Using diode laser as an activator Regarding tooth whitening and color stability 1 Day , 1 weeks, 1 month after treatment using Vita easy shade.

ELIGIBILITY:
Inclusion Criteria:

* discolored crown, non-vital or endodontically treated upper central and lateral incisors
* previous endodontic treatment performed two or more years earlier.

Exclusion Criteria:

* caries on upper central and lateral incisors, inadequate fillings, and progressive periodontal disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Color change | these assessments were performed for 1 day, 1 week, and 1 month after treatment with Vita easy shade.
  these assessments were performed for 1 day, 1 week, and 1 month after treatment with Vita easy shade obtaining difference ∆E* values using colorcoordinates CIE L*, a* and b*
color change using digital vita easy shade guide | 1 day , 1 week , 1 month
  color change using digital vita easy shade guide

CONTACTS AND LOCATIONS:
Overall Officials: Manal abd el baky A dr, phd, Study Director — Lecturer in conservative surgery departement
Locations (1):
- Misr University for science and technology, Giza, Egypt, Egypt